CLINICAL TRIAL: NCT04211077
Title: Suicidal Risk Factors Associated With Opioid Analgesics Use : a Pharmacoepidemiological Study
Brief Title: Suicidal Risk Factors Associated With Opioid Analgesics Use
Acronym: SANTE
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Collaborators: CHU Clermont Ferrand - Dpt Pharmacologie Médicale (Pr Nicolas AUTHIER) (Unknown)
Responsible Party: Sponsor
Other Study IDs: RECHMPL18_0428
Record Dates: First submitted 2019-12-18; First posted 2019-12-26 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-09

CONDITIONS: SNIIRAM Database
Keywords: Suicide attempt; Analgesics; Opioid; pharmacoepiemiology
MeSH Terms: conditions — Suicide, Attempted

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: Occurrence of a SA according to PMSI
  Interventions: Other: Date collection
- Group 2: Occurrence of accidental opioid analgesics overdose according to PMSI code
  Interventions: Other: Date collection
- Group 3: Controls : Absence of SA and accidental opioid analgesics overdose
  Interventions: Other: Date collection

INTERVENTIONS:
Other: Date collection — Data collection from national SNIIRAM and PMSI database

SUMMARY:
There is an increase in prescriptions for analgesics opioids and overdose mortality in France.

In the United States, the consumption of opioid analgesics is associated with excess mortality, especially suicide. In France, the investigator team showed retrospectively a link between history of suicide attempt (SA) and use of analgesics in general elderly population.

It is important to determine if there is a link between the prescription of opioid analgesics and suicide attempts, in a longitudinal study in general population.

The originality of the project lies in:

* the absence of a French epidemiological study on the link between opioid analgesics and suicide attempt / mortality despite the context of "opioid crisis",
* taking into account the terms of consumption of care

DETAILED DESCRIPTION:
Main objective:

To estimate the relative risk (Odds ratio) of SA associated with exposure to opioid analgesics in a case-crossover design study

Secondary objectives:

1. To Compare the profile of subjects who attempted suicide versus subjects who had an accidental drug intoxication with opioids vs subjects who did not attempt suicide or did not have an accidental overdose with opioid analgesics (case-control design)
2. To Evaluate the dose-effect of opioid analgesics on the risk of SA (case-control and case-crossover design).
3. To Identify changes in care consumption (medical consultations, co-prescriptions, changes in analgesic doses) in the 3 months preceding a SA in patients who received at least one prescription for opioid analgesics in the same period.

The Database is retrospective (2012-2017) Two methods will be used

-case crossover study (reference period of 3 months preceding the SA versus 3 control periods of 3 months without SA.- Case control study (Age and gender matching) Case 1 = occurrence of a SA according to PMSI codes "X60 to X84" between the date of the first delivery of opioid analgesics recorded in the SNIIRAM database since 2012 and December 2017; Case 2 = subjects who had accidental drug intoxication with opioid analgesics according to PMSI code "T40"; Controls = absence of SA and accidental opioid overdose

ELIGIBILITY:
Inclusion criteria:

* adults >18 years
* having received at least one reimbursed delivery of an opioid analgesic (morphine, oxycodone, fentanyl, tramadol, codeine, or lamaline) over the period 2012-2017 (SNIIRAM database).

Exclusion criteria:

- refund of methadone or buprenorphine over the period 2012-2017 (SNIIRAM database).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: having received at least one reimbursed delivery of an opioid analgesic (morphine, oxycodone, fentanyl, tramadol, codeine, or lamaline) but who have never received a refund of methadone or buprenorphine over the period 2012-2017 (SNIIRAM database).
Sampling Method: Non-Probability Sample
Enrollment: 273221 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Suicidal Risk Factors Associated with Opioid Analgesics Use | 1 year
  Occurrence of a suicide attempt

SECONDARY OUTCOMES:
Socio-demographic characteristics (potential risk factor) | 1 year
  age, gender, socioeconomical status
Other analgesic use (potential risk factor) | 1 year
  Prescription of opioid and non-opioid analgesics (name, duration of prescription, average daily dose)
Psychotropic use (potential risk factor) | 1 year
  Prescription psychotropic drugs (name, duration of prescription, average daily dose)
Comorbidities (potential risk factor) | 1 year
  Presence of somatic and psychiatric comorbidities
Care consumption (potential risk factor) | 1 year
  number, frequency and duration of hospitalizations, number and frequency of consultations (general practitioner, psychiatrist)
Nomadism indicator (potential risk factor) | 1 year
  nomadism indicator (proportion of drugs obtained with overlapping prescriptions and from different doctors over all reimbursed quantities)
Delay between first prescription of opioid analgesics and occurrence of suicide attempt | 1 year
  delay between first prescription of opioid analgesics and occurrence of suicide attempt

CONTACTS AND LOCATIONS:
Overall Officials: Emile OLIE, MD, PhD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC

REFERENCES:
- [Derived] Nobile B, Nogue E, Picot MC, Courtet P, Chenaf C, Authier N, Olie E. Association Between Opioid Analgesics and Suicide Attempts: A Nationwide French Case-Crossover Study. CNS Drugs. 2025 Dec;39(12):1331-1340. doi: 10.1007/s40263-025-01221-4. Epub 2025 Aug 30. PMID 40884605